CLINICAL TRIAL: NCT00074230
Title: Vaccination of Stage IV Cutaneous Melanoma Patients With Mature, Autologous Monocyte-Derived Dendritic Cells Transfected With RNAs Encoding for Mage-3, MelanA, and Survivin Antigens
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Cutaneous Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, PD Dr. med. univ. Beatrice Schuler-Thurner, Principal Investigator, University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERLANGEN-DERMA-ER-DC-06; CDR0000343699 (Registry Identifier: PDQ (Physician Data Query)); EU-20317
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MAGEA3 protein, human; MART-1 Antigen; Survivin

INTERVENTIONS:
Biological: Autologous Dendritic Cells loaded with MAGE-A3, MelanA and Survivin — Within cohort 1 patients received the vaccine intradermally; in cohort 2 the route of Administration was intravenous Infusion, half of the patients had additional loading with RNA coding for EL-Selektin; in cohort 3 the vaccines was again infused intravenously, the cells were matured not with MCM.mimic as in cohort 1 and 2 but either with TriMix or MCM-mimic plus CD40L-RNA.

SUMMARY:
RATIONALE: Vaccines made from a person's dendritic cells and antigens may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy using autologous dendritic cells with antigens in treating patients who have stage IV cutaneous melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of vaccination with autologous monocyte-derived dendritic cells (DC) transfected with RNAs encoding Melan-A, MAGE-3, and survivin antigens in patients with stage IV cutaneous melanoma.
* Determine whether tumor antigen-specific T-cell responses are induced in patients treated with this vaccine.
* Determine whether simultaneous loading of DC with keyhole limpet hemocyanin (KLH) significantly enhances induction of the Melan-A, MAGE-3, and survivin antigens in these patients.

Secondary

* Determine clinical antitumor activity (e.g., objective tumor response, time to tumor progression, progression-free interval, and overall survival) in patients treated with this vaccine.

OUTLINE: This is an open-label, nonrandomized study.

* Phase I: Beginning 9-11 days before vaccination, patients undergo leukapheresis for collection of peripheral blood mononuclear cells (PBMCs). PBMCs are processed for the generation of dendritic cells (DC) to be used for vaccinations. PBMCs are transfected with RNAs encoding for Melan-A, MAGE-3, and survivin antigens. DC are pulsed with keyhole limpet hemocyanin (KLH) for some patients.

Patients receive antigen-pulsed (with or without KLH) DC vaccination subcutaneously (SC) on days 1, 15, 43, and 71 in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may proceed to the phase II portion of the study.

* Phase II: Patients undergo leukapheresis as in phase I on days 102, 354, and 690. Patients receive up to 6 additional booster vaccinations SC as in phase I on days 127, 185, 269, 356, 521, and 692.

Patients are followed for 10 years.

PROJECTED ACCRUAL: A total of 8-30 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous* melanoma

  * Stage IV
* Incurable by surgical resection
* Progressive disease after at least 1 standard chemotherapy or chemoimmunotherapy regimen (e.g., dacarbazine or cisplatin monotherapy)
* Unidimensionally or bidimensionally measurable disease by physical examination (e.g., cutaneous metastases) and/or noninvasive radiological procedures
* No active CNS metastases by CT scan or MRI

  * Previously treated (e.g., excision of a single metastasis) CNS metastases are allowed provided there are no signs of active CNS metastases NOTE: *Metastatic melanoma with unidentified primary tumor allowed provided an ocular melanoma can be definitely excluded and origin from the skin is likely

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 4 months

Hematopoietic

* WBC greater than 2,500/mm^3
* Neutrophil count greater than 1,000/mm^3
* Lymphocyte count greater than 700/mm^3
* Platelet count greater than 75,000/mm^3
* Hemoglobin greater than 9 g/dL
* No bleeding disorder

Hepatic

* Bilirubin less than 2.0 mg/dL
* No evidence of hepatitis B or C infection

Renal

* Creatinine less than 2.5 mg/dL

Cardiovascular

* No clinically significant heart disease

Pulmonary

* No respiratory disease

Immunologic

* HIV-1 and HIV-2 negative
* HTLV-1 negative
* No active systemic infection
* No immunodeficiency disease
* No active autoimmune disease (e.g., lupus erythematosus, autoimmune thyroiditis or uveitis, multiple sclerosis, or inflammatory bowel disease)

  * Vitiligo allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 weeks after study participation
* Stable medical condition
* No other major serious illness
* No contraindication to leukapheresis
* No organic brain syndrome or significant psychiatric abnormality that would preclude study participation or follow-up
* No other active malignant neoplasm

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy
* No other concurrent immunotherapy during and for 2 weeks after study participation

Chemotherapy

* More than 4 weeks since prior systemic chemotherapy (6 weeks for nitrosoureas [e.g., fotemustine])
* No concurrent chemotherapy during and for 2 weeks after study participation

Endocrine therapy

* No concurrent corticosteroids during and for 2 weeks after study participation

Radiotherapy

* More than 2 weeks since prior radiotherapy
* No prior radiotherapy to the spleen
* Concurrent palliative radiotherapy to selected metastases (e.g., due to pain or local complications such as compression) is allowed

Surgery

* Recovered from prior surgery
* No prior splenectomy
* No prior organ allografts
* Concurrent surgical therapy to selected metastases (e.g., due to pain or local complications such as compression) is allowed

  * Selected accessible metastases may be removed for tumor infiltrating lymphocyte assay or other immunomonitoring investigations (e.g., expression of tumor antigens and HLA molecules)

Other

* No other concurrent investigational drug or paramedical substance during and for 2 weeks after study participation
* No concurrent participation in another clinical trial
* Concurrent palliative medication allowed (e.g., acetaminophen, indomethacin, or opiates)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability at every visit | 3 months
Overall survival as assessed by clinical staging (CT scan, positron emission tomography [PET]) every 3 months | 3 months

SECONDARY OUTCOMES:
Time to progression as assessed by clinical staging (CT scan, PET) every 3 months | 3 months
Objective tumor response as assessed by clinical staging (CT scan, PET) every 3 months | 3 months
Duration of response as assessed by clinical staging (CT scan, PET) every 3 months | 3 months
Induction of antigen-specific immune responses as assessed by elispot and tetramer staining at every visit | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Schuler, Principal Investigator — Dermatologische Klinik MIT Poliklinik-Universitaetsklinikum Erlangen
Locations (1):
- Dermatologische Klinik mit Poliklinik - Universitaetsklinikum Erlangen, Erlangen, Germany